CLINICAL TRIAL: NCT00003413
Title: High Dose Chemotherapy With Stem Cell Rescue in Recently Diagnosed Patients With Advanced (Stage III and IV) Ovarian Cancer With > 1 cm Residual Disease After Debulking Surgery
Brief Title: Combination Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Stage III or Stage IV Ovarian Epithelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Maryland Greenebaum Cancer Center (Other)
Responsible Party: UM Greenebaum Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000066426; MSGCC-9749; NCI-V98-1452
Record Dates: First submitted 1999-11-01; First posted 2004-08-03 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Ovarian Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Filgrastim; Carmustine; Cisplatin; Melphalan; Paclitaxel; Peripheral Blood Stem Cell Transplantation; Surgical Procedures, Operative

INTERVENTIONS:
Biological: filgrastim
Drug: carmustine
Drug: cisplatin
Drug: melphalan
Drug: paclitaxel
Procedure: peripheral blood stem cell transplantation
Procedure: surgical procedure

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus peripheral stem cell transplantation in treating patients with stage III or stage IV ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the complete response rates, event free survival, and overall survival of patients with recently diagnosed stage III or IV ovarian epithelial cancer receiving carmustine plus melphalan followed by consolidation therapy after having undergone surgical debulking. II. Evaluate the therapy related mortality associated with the autotransplant and the consolidation therapy in these patients. III. Evaluate the quality of life in this patient population.

OUTLINE: Patients are stratified by stage (III vs IV) and volume of residual disease (less than 3 cm vs at least 3 cm). Approximately 10-15 days after surgery, patients receive filgrastim (G-CSF) subcutaneously daily until all peripheral blood stem cell (PBSC) collections have been completed. Patients then receive carmustine IV over 2 hours on day -2 and melphalan IV over 20 minutes on day -1. Peripheral blood stem cells are infused 24 hours after melphalan on day 0. Patients receive G-CSF subcutaneously beginning on day 6 and continuing until granulocytes have recovered. Three months after the PBSC infusion, patients receive consolidation therapy with paclitaxel IV over 6 hours on day 2 and cisplatin IV over 24 hours on day 3. Consolidation treatment is repeated every 3 months for a total of 4 courses. Quality of life questionnaires are completed prior to PBSC transplant, before discharge after transplant, before each consolidation treatment, and 3 months after the last consolidation course. Patients are followed at least every 3 months for the first 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: An estimated 32 patients will be accrued into this study over 3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage III or IV ovarian epithelial cancer who have undergone surgical debulking Stage III patients must have greater than 1 cm residual mass after surgery Must have had no more than 1 course of platinum based chemotherapy No CNS disease

PATIENT CHARACTERISTICS: Age: 18 to 70 Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 1.5 mg/dL Transaminases no greater than 4 times upper limit of normal No active chronic hepatitis or liver cirrhosis Renal: Creatinine no greater than 3.0 mg/dL Cardiovascular: LVEF at least 50% Pulmonary: FVC, FEV1, and corrected DLCO at least 50% of predicted If unable to complete pulmonary function tests due to pain related to the recent surgery, patient must have a high resolution CT scan of the chest and acceptable arterial blood gases (PO2 at least 70) Other: HIV negative No active infection requiring intravenous antibiotics Not pregnant or nursing Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 1998-09; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra E. Brooks, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (1):
- Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland, United States